CLINICAL TRIAL: NCT05575466
Title: Thromboembolism in Anorexia Nervosa: a Registry-based Study of a National Cohort and a Case-control Study of the Hemostatic Balance and Its Association with Nutritional Status, Insulin and Cortisol
Brief Title: Thromboembolism in Anorexia Nervosa
Acronym: TEAN
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jeanie Meincke Egedal, MD, Medical Doctor, Odense University Hospital
Other Study IDs: 85860
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Anorexia Nervosa; Thrombosis; Thromboembolism
Keywords: Anorexia Nervosa; Thrombosis; Thromboembolism; Cortisol; Insulin; Nutrition; Refeeding Syndrome
MeSH Terms: conditions — Anorexia Nervosa; Thrombosis; Thromboembolism; Insulin Resistance; Refeeding Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Will have thromboembolic incidence rate evaluated and will have a battery of hemostatic markers analyzed
  Interventions: Diagnostic Test: Blood samples; Diagnostic Test: Questionnaires
- Controls: Will have thromboembolic incidence rate evaluated and will have a battery of hemostatic markers analyzed
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — Hemostatic biomarkers
Diagnostic Test: Questionnaires — Eating Disorder Inventory - third version (EDI-3) Eating Disorder Quality of Life Scale (EDQLS)
  Groups: Patients

SUMMARY:
BACKGROUND: Sudden death due to thromboembolic (TE) events in patients with anorexia nervosa (AN) is well known. However, the incidence of TE events and the hemostatic balance in patients with AN are sparsely investigated. Also, associations between re-nutrition and the hemostatic balance have not been studied.

OBJECTIVE: To describe the incidence of TE events in patients with AN compared to the background population, to characterize the hemostatic balance in AN compared to normal-weight women, and to assess the associations between the hemostatic balance and nutritional status, insulin sensitivity and cortisol level in women with AN.

METHODS: The incidence of TE will be described using a Danish cohort of AN patients (n=10,049) with follow-up in national registries. A comprehensive battery of hemostatic biomarkers will be compared in a case-control study of 40 patients with AN and associations between hemostasis and nutritional status will be studied.

DETAILED DESCRIPTION:
BACKGROUND

Anorexia nervosa (AN) is a complex psychiatric disorder with concomitant medical complications to malnutrition and starvation and it is associated with the highest mortality of the mental illnesses.

It is estimated that one-third of all deaths in patients with AN are due to cardiac causes, mainly sudden death, and alterations in cardiac electrical activity, structure and hemodynamics have been suggested as mortality causes. Thrombotic disorders such as myocardial infarction, stroke, and pulmonary embolism may also result in sudden cardiac death, and the investigators have previously reported venous thromboembolism in four patients with AN

Whether a disturbed hemostatic balance is associated with re-nutrition, insulin sensitivity and cortisol in AN is unknown. The guidelines of thromboprophylaxis treatment may not be appropriate in this patient group due to metabolic and hemostatic disturbances and increased thrombotic risk of reasons related to refeeding syndrome not listed in current guidelines. To optimize guidelines for AN patients, new evidence is highly warranted

AIMS

This study aims to determine the incidence of venous and arterial thromboembolic events in patients with AN compared to the background population, to characterize the hemostatic balance in AN compared to normal-weight women, and to assess the associations between the hemostatic balance and nutritional status, insulin sensitivity and cortisol level in women with AN. The study will provide new knowledge which qualifies the work of preparing guidelines for thrombosis prophylactic intervention in this patient group.

RESEARCH QUESTIONS

1. Is the incidence of venous and arterial thromboembolism increased in patients diagnosed with AN compared to an age-matched control group?
2. Is the hemostatic balance disturbed in women with AN compared with healthy, normal-weight women?
3. Are cortisol, insulin sensitivity and nutritional status associated with alterations in biomarkers of the hemostatic balance in AN?

The research questions will be answered in three sub studies.

SUB STUDY 1

Sub study 1 will answer research question 1, determining if the incidence of venous and arterial thromboembolism is increased in patients with AN compared to an age-matched control group. The study is based on the comprehensive Danish registries. An already existing cohort of more than 10,000 patients with AN will be evaluated for incidence of thromboembolic events and compared to an age-matched control group.

SUB STUDY 2

Sub study 2 will answer research question 2, exploring the hemostatic balance in patients with AN compared to healthy, normal-weight controls.

Patients with anorexia nervosa (n=40) will be recruited from the highly specialized Center of Eating Disorders at Odense University Hospital. Patients and controls will have blood samples drawn to evaluate the hemostatic balance using a large battery of hemostatic markers.

SUB STUDY 3

Sub study 3 will answer research question 3, clarifying associations between the hemostatic balance and cortisol, insulin sensitivity and nutritional status in AN. Participants of sub study 3 are the patients with AN from sub study 2. From further analysis of the blood samples and by answering validated questionnaires to determine nutritional status and AN severity, research question 3 will be answered.

ELIGIBILITY:
Inclusion Criteria, patients:

* Fulfilling Diagnostic and Statistical Manual V (DSM-5) criteria for AN
* Age 18 - 50 years
* Female sex

Exclusion Criteria, patients:

* Somatic comorbidity requiring systemic medications
* Previous thromboembolic event and/or known genetic predisposition
* Use of p.o. hormonal contraception
* Smoking

Inclusion Criteria, controls:

* BMI 18.5 - 25.0
* Age 18 - 50 years
* Female sex

Exclusion Criteria, controls:

* Somatic comorbidity requiring systemic medications
* Previous thromboembolic event and/or known genetic predisposition
* Use of p.o. hormonal contraception
* Smoking

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with anorexia nervosa and healthy, age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of thromboembolic events | Data on thromboembolic events are collected from health registries. Data is collected through study completion of the time frame in the registry, up to 26 years.
  Arterial and venous thrombosis. Non-fatal outcomes of a thromboembolic event will be validated by the use of anticoagulants in the period immediately after the outcome defining event.

OTHER OUTCOMES:
Hemostatic balance | The study is cross-sectional. Time frame for completion of participation in the study is 1 day.
  Evaluation of differences of measurements of hemostatic biomarkers in patients with AN compared to healthy controls.
  Hemostatic biomarkers that will be evaluated:
  Tissue factor TF:Ag, pg/mL
  Contact activation (descriptive, system is assessed)
  Fibrinogen mg/dl
  Thrombin generation (descriptive)
  Prothrombin fragment 1+2 pmol/L
  Plasminogen activator inhibitor type 1 ng/mL
  Tissue plasminogen activator ng/mL
  Fibrin clot properties (descriptive, using turbidity measurements)
Rotational Thromboelastometry (ROTEM)-variables | The study is cross-sectional. Time frame for completion of participation in the study is 1 day.
  Evaluation of differences in ROTEM-variables in patients with AN compared to healthy controls.

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (4):
  - Clinical Pharmacology and Pharmacy, University of Southern Denmark, Odense, Fyn
  - Department of Child and Adolescent Mental Health Odense, Mental Health Services in the Region of Southern Denmark, Odense, Fyn
  - The Nutritional Unit, Department of Endocrinology, Center for Eating Disorders, Odense University Hospital and Psychiatry in the region of Southern Denmark, Odense, Fyn
  - Unit for Thrombosis Research, Department of Clinical Biochemistry, Hospital of South West Jutland, Esbjerg, Jylland
- Department of Clinical Sciences, Umeå University, Umeå, Västerbotten County, Sweden